CLINICAL TRIAL: NCT02433340
Title: Phase 2, Multicenter, Open-Label Extension (OLE) Study With ABT-122 in Rheumatoid Arthritis Subjects Who Have Completed the Preceding M12-963 Phase 2 Randomized Controlled Trial (RCT)
Brief Title: Phase 2, Multicenter, Open-Label Extension Study With ABT-122 in Rheumatoid Arthritis Subjects Who Have Completed the Preceding M12-963 Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M12-965; 2014-001471-31 (EudraCT Number)
Record Dates: First submitted 2015-04-02; First posted 2015-05-05 (Estimated); Results first posted 2017-06-19 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Tolerability; Methotrexate; Safety
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ABT-122

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ABT-122 120 mg EOW (Experimental): All subjects receive open-label ABT-122 120 mg EOW subcutaneously, with the first dose administered at the last visit of Study M12-963 randomized controlled trial.
  Interventions: Drug: ABT-122

INTERVENTIONS:
Drug: ABT-122
  Other Names: Remtolumab

SUMMARY:
This is a Phase 2, multicenter, 24-week OLE study to assess the safety and tolerability of ABT-122 in participants with rheumatoid arthritis (RA) who had had an inadequate response to methotrexate (MTX) therapy and who completed the preceding Study M12-963 randomized controlled trial, in which participants had been randomized to receive 1 of 3 doses of ABT-122 (60 mg every other week [EOW], 120 mg EOW, or 120 mg every week [EW]) or adalimumab 40 mg EOW given on background methotrexate.

ELIGIBILITY:
Inclusion Criteria: - Subjects who have completed the preceding Study M12-963 (ABT-122) randomized controlled study and have not developed any discontinuation criteria, as defined in Study M12-963.

* If female, subject must meet one of the following criteria:

  1. Postmenopausal (defined as no menses for at least 1 year).
  2. Surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy).
  3. Practicing appropriate birth control, from the time of enrollment in this study until at least 150 days after the last dose of study drug.
* Male who agrees to follow one of the protocol-specified pregnancy avoidance measures, including refraining from donating sperm, for up to 150 days post last dose of study drug.
* Subjects must voluntarily sign and date an informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.
* Subject is judged to be in good health as determined by the Investigator based on the results of medical history, physical examination and laboratory profile performed.

Exclusion Criteria: - Pregnant or breastfeeding female.

* Ongoing infections at Day 1 (Week 0) that have NOT been successfully treated within 14 days.
* Anticipated requirement or receipt of any live vaccine during study participation including up to 120 days after the last dose of study drug.
* Current enrollment in another investigational study; with the exception of Study M12-963, which is required.
* Consideration by the Investigator, for any reason, that the subject is an unsuitable candidate to receive ABT-122.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Peloso, MD, Study Director — AbbVie

REFERENCES:
- [Derived] Khatri A, Klunder B, Peloso PM, Othman AA. Exposure-response analyses demonstrate no evidence of interleukin 17A contribution to efficacy of ABT-122 in rheumatoid or psoriatic arthritis. Rheumatology (Oxford). 2019 Feb 1;58(2):352-360. doi: 10.1093/rheumatology/key312. PMID 30376130
- [Derived] Genovese MC, Weinblatt ME, Mease PJ, Aelion JA, Peloso PM, Chen K, Li Y, Liu J, Othman AA, Khatri A, Mansikka HT, Leszczynski P. Dual inhibition of tumour necrosis factor and interleukin-17A with ABT-122: open-label long-term extension studies in rheumatoid arthritis or psoriatic arthritis. Rheumatology (Oxford). 2018 Nov 1;57(11):1972-1981. doi: 10.1093/rheumatology/key173. PMID 30032191

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 158 participants (98% of those eligible) diagnosed with active rheumatoid arthritis (RA) on background methotrexate who had participated in the randomized controlled trial M12-963 (NCT02141997) enrolled in this open-label extension. Results include analyses of data for these participants from time points during M12-963, per protocol.
Groups:
- ADA 40 mg EOW / ABT-122 120 mg EOW: Double-blind Adalimumab (ADA) 40 mg every other week (EOW) for 11 weeks. Open-label ABT-122 120 mg EOW.
- ABT-122 60 mg EOW / 120 mg EOW: Double-blind ABT-122 60 mg EOW for 11 weeks. Open-label ABT-122 120 mg EOW.
- ABT-122 120 mg EOW / 120 mg EOW: Double-blind ABT-122 120 mg EOW for 11 weeks. Open-label ABT-122 120 mg EOW.
- ABT-122 120 mg EW / 120 mg EOW: Double-blind ABT-122 120 mg every week (EW) for 11 weeks. Open-label ABT-122 120 mg EOW.
Period: Overall Study
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW
Started | 42 | 37 | 39 | 40
Completed | 40 | 35 | 37 | 38
Not Completed | 2 | 2 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Required Alternative/Prohibited Therapy | 1 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ADA 40 mg EOW / ABT-122 120 mg EOW: Double-blind ADA 40 mg EOW for 11 weeks. Open-label ABT-122 120 mg EOW.
- Total: Total of all reporting groups
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | Total
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 4 | 5 | 7 | 5 | 21
  40 to < 65 years | 27 | 24 | 22 | 26 | 99
  >= 65 years | 11 | 8 | 10 | 9 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 29 | 33 | 32 | 124
  Male | 12 | 8 | 6 | 8 | 34

OUTCOME MEASURES:

1. Primary Outcome: American College of Rheumatology (ACR) 20 Response Rate at Week 2
Description: Percentage of participants with an ACR20 response, defined as at least 20% reduction (improvement) compared with baseline in tender joint count (TJC68), swollen joint count (SJC66), and at least 3 of the 5 remaining ACR core set measures: patient's assessment of pain, patient's global assessment of disease activity (PtGA); physician's global assessment of disease activity (PGA), Health Assessment Questionnaire - Disability Index (HAQ-DI), and high-sensitivity C-reactive protein (hsCRP). Estimates of the 95% confidence interval of the response rates for each treatment group were calculated using the Agrestil-Coull method.
Time Frame: Week 2 of Study M12-963
Population: Safety Analysis Set: all participants who received at least 1 dose of study medication in M12-965 and had an assessment. Last observation carried forward (LOCF) was used for missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- All ABT-122 120 mg EOW: Open-label ABT-122 120 mg EOW.
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 40 | 37 | 39 | 38 | 154
percentage of participants | 45.0 [30.7 to 60.2] | 43.2 [28.7 to 59.1] | 46.2 [31.6 to 61.4] | 47.4 [32.5 to 62.7] | 45.5 [37.8 to 53.3]

2. Primary Outcome: ACR20 Response Rate at Week 4
Description: Percentage of participants with an ACR20 response, defined as at least 20% reduction (improvement) compared with baseline in TJC68, SJC66, and at least 3 of the 5 remaining ACR core set measures: patient's assessment of pain, PtGA; PGA, HAQ-DI, and hsCRP. Estimates of the 95% confidence interval of the response rates for each treatment group were calculated using the Agrestil-Coull method.
Time Frame: Week 4 of Study M12-963
Population: Safety Analysis Set: all participants who received at least 1 dose of study medication in M12-965 and had an assessment. LOCF was used for missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 39 | 157
percentage of participants | 50.0 [35.5 to 64.5] | 64.9 [48.7 to 78.2] | 46.2 [31.6 to 61.4] | 74.4 [58.8 to 85.6] | 58.6 [50.8 to 66.0]

3. Primary Outcome: ACR20 Response Rate at Week 6
Description: as for outcome 2
Time Frame: Week 6 of Study M12-963
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 39 | 157
percentage of participants | 66.7 [51.5 to 79.1] | 70.3 [54.1 to 82.6] | 66.7 [50.9 to 79.4] | 79.5 [64.2 to 89.5] | 70.7 [63.1 to 77.3]

4. Primary Outcome: ACR20 Response Rate at Week 8
Description: as for outcome 2
Time Frame: Week 8 of Study M12-963
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
percentage of participants | 76.2 [61.3 to 86.7] | 75.7 [59.7 to 86.8] | 69.2 [53.5 to 81.5] | 80.0 [65.0 to 89.8] | 75.3 [68.0 to 81.4]

5. Primary Outcome: ACR20 Response Rate at Week 12
Description: as for outcome 2
Time Frame: Week 12 of Study M12-963 (considered Week 0 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
percentage of participants | 78.6 [63.8 to 88.5] | 70.3 [54.1 to 82.6] | 84.6 [69.9 to 93.1] | 82.5 [67.7 to 91.6] | 79.1 [72.1 to 84.8]

6. Primary Outcome: ACR20 Response Rate at Week 16
Description: as for outcome 2
Time Frame: Week 16 (Week 4 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 41 | 36 | 37 | 40 | 154
percentage of participants | 85.4 [71.2 to 93.5] | 77.8 [61.7 to 88.5] | 86.5 [71.5 to 94.6] | 77.5 [62.3 to 87.9] | 81.8 [74.9 to 87.2]

7. Primary Outcome: ACR20 Response Rate at Week 20
Description: as for outcome 2
Time Frame: Week 20 (Week 8 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 39 | 156
percentage of participants | 71.4 [56.3 to 82.9] | 77.8 [61.7 to 88.5] | 82.1 [67.0 to 91.3] | 79.5 [64.2 to 89.5] | 77.6 [70.4 to 83.4]

8. Primary Outcome: ACR20 Response Rate at Week 24
Description: as for outcome 2
Time Frame: Week 24 (Week 12 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 39 | 156
percentage of participants | 78.6 [63.8 to 88.5] | 77.8 [61.7 to 88.5] | 76.9 [61.5 to 87.6] | 84.6 [69.9 to 93.1] | 79.5 [72.4 to 85.1]

9. Primary Outcome: ACR20 Response Rate at Week 28
Description: as for outcome 2
Time Frame: Week 28 (Week 16 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 39 | 156
percentage of participants | 73.8 [58.8 to 84.8] | 75.0 [58.7 to 86.4] | 74.4 [58.8 to 85.6] | 82.1 [67.0 to 91.3] | 76.3 [69.0 to 82.3]

10. Primary Outcome: ACR20 Response Rate at Week 32
Description: as for outcome 2
Time Frame: Week 32 (Week 20 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
percentage of participants | 76.2 [61.3 to 86.7] | 72.2 [55.9 to 84.3] | 79.5 [64.2 to 89.5] | 80.0 [65.0 to 89.8] | 77.1 [69.9 to 83.0]

11. Primary Outcome: ACR20 Response Rate at Week 36
Description: as for outcome 2
Time Frame: Week 36 (Week 24 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
percentage of participants | 71.4 [56.3 to 82.9] | 72.2 [55.9 to 84.3] | 84.6 [69.9 to 93.1] | 85.0 [70.5 to 93.3] | 78.3 [71.2 to 84.1]

12. Primary Outcome: ACR50 Response Rate at Week 2
Description: Percentage of participants with an ACR50 response, defined as at least 50% reduction (improvement) compared with baseline in TJC68, SJC66, and at least 3 of the 5 remaining ACR core set measures: patient's assessment of pain, PtGA; PGA, HAQ-DI, and hsCRP. Estimates of the 95% confidence interval of the response rates for each treatment group were calculated using the Agrestil-Coull method.
Time Frame: Week 2 of Study M12-963
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 40 | 37 | 39 | 39 | 155
percentage of participants | 10.0 [3.4 to 23.6] | 8.1 [2.1 to 22.0] | 20.5 [10.5 to 35.8] | 23.1 [12.4 to 38.5] | 15.5 [10.6 to 22.1]

13. Primary Outcome: ACR50 Response Rate at Week 4
Description: as for outcome 12
Time Frame: Week 4 of Study M12-963
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 39 | 157
percentage of participants | 14.3 [6.3 to 28.2] | 29.7 [17.4 to 45.9] | 23.1 [12.4 to 38.5] | 35.9 [22.7 to 51.6] | 25.5 [19.3 to 32.8]

14. Primary Outcome: ACR50 Response Rate at Week 6
Description: as for outcome 12
Time Frame: Week 6 of Study M12-963
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
percentage of participants | 33.3 [20.9 to 48.5] | 35.1 [21.8 to 51.3] | 38.5 [24.9 to 54.1] | 42.5 [28.5 to 57.8] | 37.3 [30.2 to 45.1]

15. Primary Outcome: ACR50 Response Rate at Week 8
Description: as for outcome 12
Time Frame: Week 8 of Study M12-963
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
percentage of participants | 45.2 [31.2 to 60.1] | 29.7 [17.4 to 45.9] | 41.0 [27.1 to 56.6] | 42.5 [28.5 to 57.8] | 39.9 [32.6 to 47.7]

16. Primary Outcome: ACR50 Response Rate at Week 12
Description: as for outcome 12
Time Frame: Week 12 of Study M12-963 (considered Week 0 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 39 | 157
percentage of participants | 52.4 [37.7 to 66.6] | 37.8 [24.0 to 53.9] | 51.3 [36.2 to 66.1] | 46.2 [31.6 to 61.4] | 47.1 [39.5 to 54.9]

17. Primary Outcome: ACR50 Response Rate at Week 16
Description: as for outcome 12
Time Frame: Week 16 (Week 4 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 41 | 35 | 37 | 39 | 152
percentage of participants | 36.6 [23.5 to 51.9] | 51.4 [35.6 to 67.0] | 56.8 [40.9 to 71.3] | 56.4 [41.0 to 70.7] | 50.0 [42.1 to 57.9]

18. Primary Outcome: ACR50 Response Rate at Week 20
Description: as for outcome 12
Time Frame: Week 20 (Week 8 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
percentage of participants | 42.9 [29.1 to 57.8] | 52.8 [37.0 to 68.0] | 51.3 [36.2 to 66.1] | 52.5 [37.5 to 67.1] | 49.7 [42.0 to 57.4]

19. Primary Outcome: ACR50 Response Rate at Week 24
Description: as for outcome 12
Time Frame: Week 24 (Week 12 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 39 | 156
percentage of participants | 40.5 [27.0 to 55.5] | 47.2 [32.0 to 63.0] | 53.8 [38.6 to 68.4] | 71.8 [56.1 to 83.6] | 53.2 [45.4 to 60.9]

20. Primary Outcome: ACR50 Response Rate at Week 28
Description: as for outcome 12
Time Frame: Week 28 (Week 16 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 39 | 156
percentage of participants | 50.0 [35.5 to 64.5] | 47.2 [32.0 to 63.0] | 51.3 [36.2 to 66.1] | 69.2 [53.5 to 81.5] | 54.5 [46.7 to 62.1]

21. Primary Outcome: ACR50 Response Rate at Week 32
Description: as for outcome 12
Time Frame: Week 32 (Week 20 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
percentage of participants | 45.2 [31.2 to 60.1] | 58.3 [42.2 to 72.9] | 51.3 [36.2 to 66.1] | 62.5 [47.0 to 75.8] | 54.1 [46.3 to 61.7]

22. Primary Outcome: ACR50 Response Rate at Week 36
Description: as for outcome 12
Time Frame: Week 36 (Week 24 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
percentage of participants | 45.2 [31.2 to 60.1] | 50.0 [34.5 to 65.5] | 53.8 [38.6 to 68.4] | 62.5 [47.0 to 75.8] | 52.9 [45.1 to 60.5]

23. Primary Outcome: ACR70 Response Rate at Week 2
Description: Percentage of participants with an ACR70 response, defined as at least 70% reduction (improvement) compared with baseline in TJC68, SJC66, and at least 3 of the 5 remaining ACR core set measures: patient's assessment of pain, PtGA; PGA, HAQ-DI, and hsCRP. Estimates of the 95% confidence interval of the response rates for each treatment group were calculated using the Agrestil-Coull method.
Time Frame: Week 2 of Study M12-963
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 40 | 37 | 39 | 39 | 155
percentage of participants | 0.0 [0.0 to 10.4] | 2.7 [0.0 to 15.1] | 5.1 [0.5 to 17.8] | 5.1 [0.5 to 17.8] | 3.2 [1.2 to 7.5]

24. Primary Outcome: ACR70 Response Rate at Week 4
Description: as for outcome 23
Time Frame: Week 4 of Study M12-963
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
percentage of participants | 4.8 [0.5 to 16.6] | 10.8 [3.7 to 25.3] | 10.3 [3.5 to 24.2] | 17.5 [8.4 to 32.3] | 10.8 [6.7 to 16.6]

25. Primary Outcome: ACR70 Response Rate at Week 6
Description: as for outcome 23
Time Frame: Week 6 of Study M12-963
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
percentage of participants | 16.7 [8.0 to 30.9] | 13.5 [5.4 to 28.5] | 17.9 [8.7 to 33.0] | 20.0 [10.2 to 35.0] | 17.1 [12.0 to 23.8]

26. Primary Outcome: ACR70 Response Rate at Week 8
Description: as for outcome 23
Time Frame: Week 8 of Study M12-963
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
percentage of participants | 19.0 [9.7 to 33.6] | 8.1 [2.1 to 22.0] | 25.6 [14.4 to 41.2] | 27.5 [16.0 to 43.0] | 20.3 [14.7 to 27.2]

27. Primary Outcome: ACR70 Response Rate at Week 12
Description: as for outcome 23
Time Frame: Week 12 of Study M12-963 (considered Week 0 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
percentage of participants | 23.8 [13.3 to 38.7] | 24.3 [13.2 to 40.3] | 20.5 [10.5 to 35.8] | 35.0 [22.1 to 50.5] | 25.9 [19.7 to 33.3]

28. Primary Outcome: ACR70 Response Rate at Week 16
Description: as for outcome 23
Time Frame: Week 16 (Week 4 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 40 | 36 | 36 | 39 | 151
percentage of participants | 15.0 [6.7 to 29.5] | 30.6 [17.9 to 47.0] | 33.3 [20.1 to 49.7] | 25.6 [14.4 to 41.2] | 25.8 [19.5 to 33.4]

29. Primary Outcome: ACR70 Response Rate at Week 20
Description: as for outcome 23
Time Frame: Week 20 (Week 8 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 35 | 39 | 40 | 156
percentage of participants | 19.0 [9.7 to 33.6] | 31.4 [18.4 to 48.1] | 33.3 [20.6 to 49.1] | 32.5 [20.0 to 48.1] | 28.8 [22.3 to 36.4]

30. Primary Outcome: ACR70 Response Rate at Week 24
Description: as for outcome 23
Time Frame: Week 24 (Week 12 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
percentage of participants | 19.0 [9.7 to 33.6] | 25.0 [13.6 to 41.3] | 28.2 [16.4 to 43.9] | 40.0 [26.3 to 55.4] | 28.0 [21.6 to 35.5]

31. Primary Outcome: ACR70 Response Rate at Week 28
Description: as for outcome 23
Time Frame: Week 28 (Week 16 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 39 | 156
percentage of participants | 16.7 [8.0 to 30.9] | 27.8 [15.7 to 44.1] | 30.8 [18.5 to 46.5] | 41.0 [27.1 to 56.6] | 28.8 [22.3 to 36.4]

32. Primary Outcome: ACR70 Response Rate at Week 32
Description: as for outcome 23
Time Frame: Week 32 (Week 20 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
percentage of participants | 16.7 [8.0 to 30.9] | 27.8 [15.7 to 44.1] | 23.1 [12.4 to 38.5] | 42.5 [28.5 to 57.8] | 27.4 [21.0 to 34.9]

33. Primary Outcome: ACR70 Response Rate at Week 36
Description: as for outcome 23
Time Frame: Week 36 (Week 24 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
percentage of participants | 23.8 [13.3 to 38.7] | 30.6 [17.9 to 47.0] | 35.9 [22.7 to 51.6] | 45.0 [30.7 to 60.2] | 33.8 [26.8 to 41.5]

34. Primary Outcome: Summary of Treatment-Emergent Adverse Events (AEs), Serious AEs (SAEs), AEs Leading to Discontinuation, and Deaths
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related. An SAE is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent events (TEAEs/TESAEs) are defined as any event that began or worsened in severity after the first dose of study drug. For more details on adverse events please see the Adverse Event section.
Time Frame: from the first dose of study drug in study M12-965 until 70 days after the last dose of study drug (up to 32 weeks)
Population: Safety Analysis Set: all participants who received at least 1 dose of study medication in M12-965.
Measure: Count of Participants; unit: Participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
Participants
  Any AE | 17 | 15 | 19 | 14 | 65
  AE possibly study drug-related | 5 | 6 | 6 | 6 | 23
  SAE possibly study drug-related | 0 | 0 | 0 | 0 | 0
  Severe AE | 0 | 1 | 1 | 0 | 2
  SAE | 0 | 1 | 5 | 0 | 6
  AE leading to study drug discontinuation | 1 | 0 | 1 | 0 | 2
  AE leading to Death | 0 | 0 | 0 | 0 | 0
  Death (includes non-treatment-emergent) | 0 | 0 | 0 | 0 | 0

35. Secondary Outcome: Change From Baseline In Tender Joint Count (TJC68) at Week 2
Description: At each study visit, a joint evaluator assessed whether a particular joint was "tender or painful" where presence of tenderness was scored as "1" and the absence of tenderness was scored as "0," provided the joint was not replaced or could not be assessed due to other reasons. The total TJC68, which is based on 68 joints, was derived as the sum of all "1s" thus collected with no penalty considered for the joints not assessed or those which had been replaced. The range for TJC68 was 0 to 68, with a higher score indication a greater degree of tenderness. For analysis purposes, all baseline values are defined as the last measurement on or before the first dose of study drug in Study M12-963.
Time Frame: Week 2 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 40 | 36 | 39 | 40 | 155
tender joints | -9.4 (10.28) | -11.6 (10.57) | -11.0 (11.12) | -12.9 (13.84) | -11.2 (11.52)

36. Secondary Outcome: Change From Baseline in TJC68 at Week 4
Description: as for outcome 35
Time Frame: Week 4 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
tender joints | -13.1 (9.98) | -16.6 (12.48) | -13.6 (12.00) | -16.1 (12.77) | -14.8 (11.80)

37. Secondary Outcome: Change From Baseline in TJC68 at Week 6
Description: as for outcome 35
Time Frame: Week 6 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
tender joints | -15.8 (10.18) | -16.9 (11.67) | -15.3 (11.05) | -16.6 (12.56) | -16.1 (11.28)

38. Secondary Outcome: Change From Baseline in TJC68 at Week 8
Description: as for outcome 35
Time Frame: Week 8 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
tender joints | -17.3 (9.93) | -17.4 (10.85) | -17.1 (10.21) | -17.1 (13.33) | -17.2 (11.05)

39. Secondary Outcome: Change From Baseline in TJC68 at Week 12
Description: as for outcome 35
Time Frame: Week 12 of Study M12-963 (considered Week 0 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
tender joints | -18.4 (11.78) | -16.9 (10.90) | -18.6 (10.16) | -18.0 (12.64) | -18.0 (11.34)

40. Secondary Outcome: Change From Baseline in TJC68 at Week 16
Description: as for outcome 35
Time Frame: Week 16 (Week 4 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 41 | 36 | 37 | 40 | 154
tender joints | -18.3 (12.03) | -19.2 (10.57) | -17.6 (9.14) | -18.1 (12.38) | -18.3 (11.07)

41. Secondary Outcome: Change From Baseline in TJC68 at Week 20
Description: as for outcome 35
Time Frame: Week 20 (Week 8 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
tender joints | -17.6 (11.93) | -19.7 (10.60) | -17.8 (10.31) | -19.0 (11.89) | -18.5 (11.16)

42. Secondary Outcome: Change From Baseline in TJC68 at Week 24
Description: as for outcome 35
Time Frame: Week 24 (Week 12 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
tender joints | -19.3 (12.16) | -18.3 (10.27) | -17.4 (9.70) | -19.8 (12.32) | -18.7 (11.15)

43. Secondary Outcome: Change From Baseline in TJC68 at Week 28
Description: as for outcome 35
Time Frame: Week 28 (Week 16 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
tender joints | -18.2 (10.88) | -18.9 (12.26) | -17.9 (10.31) | -21.0 (13.02) | -19.0 (11.60)

44. Secondary Outcome: Change From Baseline in TJC68 at Week 32
Description: as for outcome 35
Time Frame: Week 32 (Week 20 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
tender joints | -18.2 (11.72) | -19.7 (11.04) | -17.9 (10.47) | -20.3 (13.38) | -19.0 (11.66)

45. Secondary Outcome: Change From Baseline in TJC68 at Week 36
Description: as for outcome 35
Time Frame: Week 36 (Week 24 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
tender joints | -18.2 (10.92) | -18.5 (11.92) | -17.7 (10.06) | -20.3 (12.88) | -18.7 (11.42)

46. Secondary Outcome: Change From Baseline in Swollen Joint Count (SJC66) at Week 2
Description: At each study visit, a joint evaluator assessed whether a particular joint was swollen where presence of swelling was scored as "1" and the absence of swelling was scored as "0," provided the joint was not replaced or could not be assessed due to other reasons. The total SJC66, which is based on 66 joints, was derived as the sum of all "1s" thus collected with no penalty considered for the joints not assessed or those which had been replaced. The range for SJC66 was 0 to 66, with a higher score indicating a greater degree of swelling. For analysis purposes, all baseline values are defined as the last measurement on or before the first dose of study drug in Study M12-963.
Time Frame: Week 2 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 40 | 36 | 39 | 40 | 155
swollen joints | -8.0 (9.07) | -8.8 (8.50) | -8.6 (10.84) | -10.8 (9.34) | -9.0 (9.46)

47. Secondary Outcome: Change From Baseline in SJC66 at Week 4
Description: as for outcome 46
Time Frame: Week 4 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
swollen joints | -8.8 (8.72) | -10.6 (8.04) | -10.3 (10.50) | -13.3 (9.29) | -10.7 (9.26)

48. Secondary Outcome: Change From Baseline in SJC66 at Week 6
Description: as for outcome 46
Time Frame: Week 6 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
swollen joints | -11.8 (8.09) | -11.9 (7.71) | -12.3 (10.15) | -13.3 (9.31) | -12.3 (8.81)

49. Secondary Outcome: Change From Baseline in SJC66 at Week 8
Description: as for outcome 46
Time Frame: Week 8 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
swollen joints | -12.2 (8.26) | -12.4 (7.76) | -13.8 (9.32) | -14.3 (9.43) | -13.2 (8.70)

50. Secondary Outcome: Change From Baseline in SJC66 at Week 12
Description: as for outcome 46
Time Frame: Week 12 of Study M12-963 (considered Week 0 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
swollen joints | -12.6 (8.73) | -11.8 (9.51) | -13.4 (9.13) | -14.8 (9.00) | -13.2 (9.06)

51. Secondary Outcome: Change From Baseline in SJC66 at Week 16
Description: as for outcome 46
Time Frame: Week 16 (Week 4 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 41 | 36 | 37 | 40 | 154
swollen joints | -13.0 (8.50) | -13.5 (9.60) | -13.8 (8.90) | -14.5 (8.69) | -13.7 (8.84)

52. Secondary Outcome: Change From Baseline in SJC66 at Week 20
Description: as for outcome 46
Time Frame: Week 20 (Week 8 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
swollen joints | -12.2 (7.47) | -14.6 (8.97) | -13.8 (10.30) | -15.4 (8.95) | -14.0 (8.95)

53. Secondary Outcome: Change From Baseline in SJC66 at Week 24
Description: as for outcome 46
Time Frame: Week 24 (Week 12 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
swollen joints | -14.0 (8.21) | -13.8 (8.68) | -14.6 (9.87) | -15.6 (9.16) | -14.5 (8.93)

54. Secondary Outcome: Change From Baseline in SJC66 at Week 28
Description: as for outcome 46
Time Frame: Week 28 (Week 16 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
swollen joints | -13.3 (6.88) | -14.0 (10.12) | -14.9 (9.49) | -15.8 (9.29) | -14.5 (8.94)

55. Secondary Outcome: Change From Baseline in SJC66 at Week 32
Description: as for outcome 46
Time Frame: Week 32 (Week 20 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
swollen joints | -13.1 (8.14) | -13.9 (10.34) | -14.3 (9.81) | -14.9 (9.71) | -14.1 (9.43)

56. Secondary Outcome: Change From Baseline in SJC66 at Week 36
Description: as for outcome 46
Time Frame: Week 36 (Week 24 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
swollen joints | -12.4 (7.76) | -14.0 (10.55) | -15.0 (9.57) | -14.8 (9.82) | -14.0 (9.40)

57. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain at Week 2
Description: Participants assessed their pain in the previous week using a Patient's Global Assessment Pain visual analogue scale (VAS). The range is 0 to 100 mm with no pain being indicated by 0 and severe pain by 100. For analysis purposes, all baseline values are defined as the last measurement on or before the first dose of study drug in Study M12-963.
Time Frame: Week 2 of Study M12-963
Population: Safety Analysis Set: all participants who received at least 1 dose of study medication in M12-965 and had a baseline and post-baseline assessment. LOCF was used for missing data; LOCF imputation was conducted separately for M12-963 and M12-965 (ie, data from M12-963 was not carried forward to visits in M12-965).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 40 | 36 | 39 | 39 | 154
units on a scale | -17.9 (22.82) | -20.1 (16.83) | -22.4 (23.49) | -22.3 (22.46) | -20.7 (21.53)

58. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain at Week 4
Description: Participants assessed their pain in the previous week using a Patient's Global Assessment Pain VAS. The range is 0 to 100 mm with no pain being indicated by 0 and severe pain by 100. For analysis purposes, all baseline values are defined as the last measurement on or before the first dose of study drug in Study M12-963.
Time Frame: Week 4 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -24.5 (20.24) | -28.7 (20.76) | -24.8 (26.57) | -29.3 (23.07) | -26.8 (22.68)

59. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain at Week 6
Description: as for outcome 58
Time Frame: Week 6 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -31.8 (21.24) | -29.1 (22.48) | -29.8 (27.07) | -29.9 (21.36) | -30.2 (22.92)

60. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain at Week 8
Description: as for outcome 58
Time Frame: Week 8 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -30.5 (24.64) | -29.8 (21.56) | -30.2 (27.89) | -36.0 (23.11) | -31.7 (24.36)

61. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain at Week 12
Description: as for outcome 58
Time Frame: Week 12 of Study M12-963 (considered Week 0 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -36.2 (19.91) | -29.3 (22.34) | -37.9 (27.18) | -36.5 (23.52) | -35.1 (23.34)

62. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain at Week 16
Description: as for outcome 58
Time Frame: Week 16 (Week 4 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 41 | 36 | 37 | 40 | 154
units on a scale | -31.9 (24.68) | -33.0 (24.11) | -35.0 (28.43) | -38.5 (22.92) | -34.6 (24.96)

63. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain at Week 20
Description: as for outcome 58
Time Frame: Week 20 (Week 8 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -30.2 (22.48) | -40.3 (24.12) | -37.8 (28.78) | -36.8 (21.72) | -36.1 (24.44)

64. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain at Week 24
Description: as for outcome 58
Time Frame: Week 24 (Week 12 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -31.7 (21.86) | -35.9 (23.28) | -32.0 (30.31) | -39.4 (23.64) | -34.7 (24.92)

65. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain at Week 28
Description: as for outcome 58
Time Frame: Week 28 (Week 16 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -28.5 (22.39) | -36.2 (28.88) | -35.3 (28.64) | -40.1 (22.61) | -34.9 (25.79)

66. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain at Week 32
Description: as for outcome 58
Time Frame: Week 32 (Week 20 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -27.3 (22.16) | -37.4 (25.63) | -34.3 (32.99) | -42.8 (25.31) | -35.3 (27.10)

67. Secondary Outcome: Change From Baseline in Patient's Assessment of Pain at Week 36
Description: as for outcome 58
Time Frame: Week 36 (Week 24 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -31.3 (23.36) | -36.1 (28.90) | -39.3 (31.37) | -41.8 (28.21) | -37.0 (28.03)

68. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity at Week 2
Description: Participants assessed their disease activity for the past 24 hours using a Patient's Global Assessment of Disease VAS. The range is 0 to 100 mm with no activity being indicated by 0 and severe activity by 100. For analysis purposes, all baseline values are defined as the last measurement on or before the first dose of study drug in Study M12-963.
Time Frame: Week 2 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 40 | 36 | 39 | 39 | 154
units on a scale | -18.1 (23.77) | -14.2 (16.41) | -21.3 (19.92) | -17.2 (23.06) | -17.7 (21.03)

69. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity at Week 4
Description: as for outcome 68
Time Frame: Week 4 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -20.6 (21.73) | -25.6 (22.33) | -20.7 (24.62) | -26.6 (21.79) | -23.3 (22.58)

70. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity at Week 6
Description: as for outcome 68
Time Frame: Week 6 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -26.5 (20.97) | -23.2 (22.21) | -26.9 (24.17) | -27.9 (21.14) | -26.2 (21.98)

71. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity at Week 8
Description: as for outcome 68
Time Frame: Week 8 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -27.1 (24.33) | -26.8 (23.25) | -31.8 (25.54) | -34.1 (22.93) | -30.0 (24.02)

72. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity at Week 12
Description: as for outcome 68
Time Frame: Week 12 of Study M12-963 (considered Week 0 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -29.2 (23.39) | -29.0 (25.11) | -34.1 (21.41) | -35.6 (25.62) | -32.0 (23.86)

73. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity at Week 16
Description: as for outcome 68
Time Frame: Week 16 (Week 4 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 41 | 36 | 37 | 40 | 154
units on a scale | -26.8 (24.09) | -29.3 (24.91) | -34.8 (20.59) | -35.8 (22.51) | -31.6 (23.18)

74. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity at Week 20
Description: as for outcome 68
Time Frame: Week 20 (Week 8 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -28.5 (20.98) | -35.6 (24.56) | -35.4 (26.44) | -35.4 (22.95) | -33.6 (23.72)

75. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity at Week 24
Description: as for outcome 68
Time Frame: Week 24 (Week 12 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -31.5 (22.81) | -33.1 (24.25) | -32.7 (25.16) | -38.9 (23.63) | -34.0 (23.89)

76. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity at Week 28
Description: as for outcome 68
Time Frame: Week 28 (Week 16 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -25.0 (23.25) | -33.1 (27.93) | -32.6 (27.33) | -39.7 (25.57) | -32.5 (26.29)

77. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity at Week 32
Description: as for outcome 68
Time Frame: Week 32 (Week 20 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -27.4 (23.87) | -34.2 (26.17) | -32.8 (28.91) | -43.8 (23.56) | -34.5 (26.12)

78. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Disease Activity at Week 36
Description: as for outcome 68
Time Frame: Week 36 (Week 24 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -29.5 (26.04) | -32.5 (26.16) | -37.5 (25.73) | -38.3 (29.65) | -34.4 (26.96)

79. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity at Week 2
Description: The physician assessed the participant's disease activity at the time of visit using a Physician's Global Assessment of Disease VAS. The range is 0 to 100 mm with no activity being indicated by 0 and severe activity by 100. For analysis purposes, all baseline values are defined as the last measurement on or before the first dose of study drug in Study M12-963.
Time Frame: Week 2 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 39 | 36 | 39 | 39 | 153
units on a scale | -24.5 (21.80) | -25.8 (17.29) | -29.5 (21.25) | -26.5 (21.54) | -26.6 (20.49)

80. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity at Week 4
Description: as for outcome 79
Time Frame: Week 4 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 39 | 156
units on a scale | -28.6 (20.49) | -35.5 (21.15) | -34.5 (21.58) | -37.3 (23.00) | -33.8 (21.61)

81. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity at Week 6
Description: as for outcome 79
Time Frame: Week 6 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 39 | 156
units on a scale | -38.5 (18.77) | -39.0 (22.76) | -40.3 (23.63) | -40.1 (20.94) | -39.5 (21.33)

82. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity at Week 8
Description: as for outcome 79
Time Frame: Week 8 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 39 | 156
units on a scale | -41.0 (17.82) | -39.6 (20.94) | -45.6 (21.16) | -43.4 (22.87) | -42.4 (20.65)

83. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity at Week 12
Description: as for outcome 79
Time Frame: Week 12 of Study M12-963 (considered Week 0 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 39 | 156
units on a scale | -44.4 (20.30) | -42.9 (20.90) | -49.7 (20.54) | -47.6 (19.86) | -46.2 (20.36)

84. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity at Week 16
Description: as for outcome 79
Time Frame: Week 16 (Week 4 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 40 | 35 | 36 | 37 | 148
units on a scale | -46.0 (17.04) | -45.3 (24.23) | -47.3 (20.99) | -47.3 (21.46) | -46.4 (20.77)

85. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity at Week 20
Description: as for outcome 79
Time Frame: Week 20 (Week 8 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 35 | 38 | 38 | 153
units on a scale | -44.3 (19.08) | -46.1 (20.28) | -45.6 (22.89) | -49.3 (21.64) | -46.3 (20.86)

86. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity at Week 24
Description: as for outcome 79
Time Frame: Week 24 (Week 12 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 39 | 156
units on a scale | -45.8 (18.06) | -46.7 (22.00) | -47.4 (23.02) | -49.9 (23.05) | -47.4 (21.40)

87. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity at Week 28
Description: as for outcome 79
Time Frame: Week 28 (Week 16 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 39 | 156
units on a scale | -44.5 (20.72) | -48.7 (22.19) | -48.2 (22.85) | -51.7 (20.85) | -48.2 (21.59)

88. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity at Week 32
Description: as for outcome 79
Time Frame: Week 32 (Week 20 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 39 | 156
units on a scale | -45.2 (23.07) | -50.0 (24.46) | -49.9 (24.42) | -51.7 (25.03) | -49.1 (24.12)

89. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity at Week 36
Description: as for outcome 79
Time Frame: Week 36 (Week 24 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 39 | 156
units on a scale | -42.4 (23.72) | -48.0 (23.10) | -50.5 (24.55) | -51.8 (24.24) | -48.1 (23.98)

90. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 2
Description: HAQ-DI is a self-reported participant outcome measurement. It is calculated as the mean of the scores from 8 following categories with a range 0 - 3: Dressing and Grooming, Rising, Eating, Walking, Hygiene, Reach, Grip, and Activities. The higher the score, the more likely to associate with morbidity and mortality for the participant. The minimum clinically important difference in HAQ-DI was defined as change from baseline ≤ -0.22. For analysis purposes, all baseline values are defined as the last measurement on or before the first dose of study drug in Study M12-963.
Time Frame: Week 2 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 40 | 36 | 39 | 39 | 154
units on a scale | -0.25 (0.486) | -0.31 (0.463) | -0.29 (0.481) | -0.40 (0.538) | -0.31 (0.492)

91. Secondary Outcome: Change From Baseline in HAQ-DI at Week 4
Description: as for outcome 90
Time Frame: Week 4 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -0.37 (0.552) | -0.40 (0.580) | -0.47 (0.625) | -0.62 (0.711) | -0.47 (0.622)

92. Secondary Outcome: Change From Baseline in HAQ-DI at Week 6
Description: as for outcome 90
Time Frame: Week 6 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -0.53 (0.601) | -0.46 (0.607) | -0.63 (0.711) | -0.64 (0.584) | -0.57 (0.626)

93. Secondary Outcome: Change From Baseline in HAQ-DI at Week 8
Description: as for outcome 90
Time Frame: Week 8 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -0.56 (0.619) | -0.52 (0.525) | -0.65 (0.648) | -0.71 (0.711) | -0.61 (0.630)

94. Secondary Outcome: Change From Baseline in HAQ-DI at Week 12
Description: as for outcome 90
Time Frame: Week 12 of Study M12-963 (considered Week 0 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -0.69 (0.654) | -0.55 (0.611) | -0.66 (0.701) | -0.88 (0.677) | -0.70 (0.667)

95. Secondary Outcome: Change From Baseline in HAQ-DI at Week 16
Description: as for outcome 90
Time Frame: Week 16 (Week 4 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 41 | 36 | 37 | 40 | 154
units on a scale | -0.59 (0.616) | -0.67 (0.631) | -0.67 (0.689) | -0.90 (0.649) | -0.71 (0.651)

96. Secondary Outcome: Change From Baseline in HAQ-DI at Week 20
Description: as for outcome 90
Time Frame: Week 20 (Week 8 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -0.54 (0.662) | -0.73 (0.555) | -0.70 (0.788) | -0.88 (0.690) | -0.71 (0.685)

97. Secondary Outcome: Change From Baseline in HAQ-DI at Week 24
Description: as for outcome 90
Time Frame: Week 24 (Week 12 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -0.63 (0.604) | -0.74 (0.617) | -0.60 (0.805) | -0.91 (0.704) | -0.72 (0.691)

98. Secondary Outcome: Change From Baseline in HAQ-DI at Week 28
Description: as for outcome 90
Time Frame: Week 28 (Week 16 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -0.60 (0.600) | -0.77 (0.630) | -0.69 (0.727) | -0.99 (0.699) | -0.76 (0.676)

99. Secondary Outcome: Change From Baseline in HAQ-DI at Week 32
Description: as for outcome 90
Time Frame: Week 32 (Week 20 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -0.54 (0.576) | -0.76 (0.674) | -0.66 (0.794) | -0.91 (0.659) | -0.71 (0.686)

100. Secondary Outcome: Change From Baseline in HAQ-DI at Week 36
Description: as for outcome 90
Time Frame: Week 36 (Week 24 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -0.62 (0.619) | -0.73 (0.698) | -0.71 (0.674) | -0.81 (0.749) | -0.72 (0.683)

101. Secondary Outcome: Change From Baseline in High-Sensitivity C-Reactive Protein (hsCRP) at Week 2
Description: For analysis purposes, all baseline are defined as the last measurement on or before the first dose of study drug in Study M12-963.
Time Frame: Week 2 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 40 | 36 | 39 | 40 | 155
mg/L | -12.6 (25.19) | -9.9 (12.89) | -12.6 (18.56) | -14.9 (25.70) | -12.5 (21.30)

102. Secondary Outcome: Change From Baseline in hsCRP at Week 4
Description: as for outcome 101
Time Frame: Week 4 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
mg/L | -13.3 (25.40) | -8.0 (12.37) | -11.7 (17.43) | -14.6 (26.51) | -12.0 (21.43)

103. Secondary Outcome: Change From Baseline in hsCRP at Week 6
Description: as for outcome 101
Time Frame: Week 6 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
mg/L | -13.3 (25.15) | -8.0 (11.98) | -10.7 (18.84) | -14.9 (26.56) | -11.8 (21.63)

104. Secondary Outcome: Change From Baseline in hsCRP at Week 8
Description: as for outcome 101
Time Frame: Week 8 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
mg/L | -12.2 (24.96) | -8.0 (13.13) | -10.7 (19.00) | -12.9 (28.42) | -11.0 (22.26)

105. Secondary Outcome: Change From Baseline in hsCRP at Week 12
Description: as for outcome 101
Time Frame: Week 12 of Study M12-963 (considered Week 0 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
mg/L | -12.3 (25.56) | -6.5 (14.05) | -10.8 (17.27) | -14.6 (25.22) | -11.2 (21.36)

106. Secondary Outcome: Change From Baseline in hsCRP at Week 16
Description: as for outcome 101
Time Frame: Week 16 (Week 4 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 41 | 36 | 37 | 39 | 153
mg/L | -13.5 (24.92) | -5.5 (17.44) | -10.8 (16.26) | -12.5 (24.65) | -10.7 (21.39)

107. Secondary Outcome: Change From Baseline in hsCRP at Week 20
Description: as for outcome 101
Time Frame: Week 20 (Week 8 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
mg/L | -11.6 (24.46) | -6.4 (14.07) | -10.3 (18.66) | -11.6 (25.06) | -10.1 (21.16)

108. Secondary Outcome: Change From Baseline in hsCRP at Week 24
Description: as for outcome 101
Time Frame: Week 24 (Week 12 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
mg/L | -11.3 (23.41) | -6.7 (13.93) | -9.1 (17.96) | -10.8 (27.79) | -9.6 (21.50)

109. Secondary Outcome: Change From Baseline in hsCRP at Week 28
Description: as for outcome 101
Time Frame: Week 28 (Week 16 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
mg/L | -3.5 (48.65) | -6.3 (17.24) | -11.3 (18.37) | -6.8 (26.24) | -6.9 (30.84)

110. Secondary Outcome: Change From Baseline in hsCRP at Week 32
Description: as for outcome 101
Time Frame: Week 32 (Week 20 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
mg/L | -9.8 (26.15) | -7.6 (14.59) | -8.0 (20.16) | -10.4 (26.24) | -9.0 (22.36)

111. Secondary Outcome: Change From Baseline in hsCRP at Week 36
Description: as for outcome 101
Time Frame: Week 36 (Week 24 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
mg/L | -8.7 (26.17) | -6.0 (16.47) | -8.7 (17.56) | -9.0 (28.55) | -8.1 (22.83)

112. Secondary Outcome: Change From Baseline in Disease Activity Score 28 (DAS28[hsCRP]) at Week 2
Description: The DAS28 (hsCRP) is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, hsCRP, and general health are included in the DAS28 (hsCRP) score. Scores range from 0 to 10, with higher scores indicating more disease activity. For analysis purposes, all baseline values are defined as the last measurement on or before the first dose of study drug in Study M12-963.
Time Frame: Week 2 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 40 | 37 | 39 | 39 | 155
units on a scale | -1.5 (1.23) | -1.5 (1.06) | -1.8 (1.27) | -1.7 (1.13) | -1.6 (1.17)

113. Secondary Outcome: Change From Baseline in DAS28 (hsCRP) at Week 4
Description: as for outcome 112
Time Frame: Week 4 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
units on a scale | -1.9 (1.20) | -2.1 (1.37) | -2.1 (1.26) | -2.3 (1.20) | -2.1 (1.25)

114. Secondary Outcome: Change From Baseline in DAS28 (hsCRP) at Week 6
Description: as for outcome 112
Time Frame: Week 6 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
units on a scale | -2.4 (1.37) | -2.2 (1.34) | -2.5 (1.27) | -2.4 (1.21) | -2.4 (1.29)

115. Secondary Outcome: Change From Baseline in DAS28 (hsCRP) at Week 8
Description: as for outcome 112
Time Frame: Week 8 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
units on a scale | -2.4 (1.29) | -2.3 (1.25) | -2.7 (1.30) | -2.6 (1.32) | -2.5 (1.28)

116. Secondary Outcome: Change From Baseline in DAS28 (hsCRP) at Week 12
Description: as for outcome 112
Time Frame: Week 12 of Study M12-963 (considered Week 0 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
units on a scale | -2.6 (1.32) | -2.3 (1.49) | -2.8 (1.17) | -2.7 (1.14) | -2.6 (1.28)

117. Secondary Outcome: Change From Baseline in DAS28 (hsCRP) at Week 16
Description: as for outcome 112
Time Frame: Week 16 (Week 4 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 41 | 36 | 37 | 39 | 153
units on a scale | -2.7 (1.21) | -2.6 (1.54) | -2.8 (1.19) | -2.6 (0.92) | -2.7 (1.22)

118. Secondary Outcome: Change From Baseline in DAS28 (hsCRP) at Week 20
Description: as for outcome 112
Time Frame: Week 20 (Week 8 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -2.7 (1.31) | -2.8 (1.37) | -2.7 (1.25) | -2.8 (1.08) | -2.7 (1.24)

119. Secondary Outcome: Change From Baseline in DAS28 (hsCRP) at Week 24
Description: as for outcome 112
Time Frame: Week 24 (Week 12 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -2.8 (1.26) | -2.6 (1.47) | -2.7 (1.41) | -2.9 (1.14) | -2.8 (1.31)

120. Secondary Outcome: Change From Baseline in DAS28 (hsCRP) at Week 28
Description: as for outcome 112
Time Frame: Week 28 (Week 16 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -2.5 (1.45) | -2.7 (1.46) | -2.9 (1.24) | -2.9 (1.06) | -2.7 (1.31)

121. Secondary Outcome: Change From Baseline in DAS28 (hsCRP) at Week 32
Description: as for outcome 112
Time Frame: Week 32 (Week 20 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -2.6 (1.44) | -2.8 (1.45) | -2.7 (1.17) | -2.9 (1.25) | -2.8 (1.32)

122. Secondary Outcome: Change From Baseline in DAS28 (hsCRP) at Week 36
Description: as for outcome 112
Time Frame: Week 36 (Week 24 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
units on a scale | -2.6 (1.45) | -2.6 (1.48) | -2.8 (1.22) | -2.8 (1.32) | -2.7 (1.36)

123. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) at Week 2
Description: CDAI is a composite index for assessing disease activity based on the summation of the counts of Tender Joint Count 28 (TJC28) and Swollen Joint Count 28 (SJC28), patient global assessment of disease activity measured on a VAS from 0 to 10 cm, and physician global assessment of disease activity measured on a VAS from 0 to 10 cm. The total CDAI score ranges from 0 to 78 with higher scores indicating higher disease activity. For analysis purposes, all baseline values are defined as the last measurement on or before the first dose of study drug in Study M12-963.
Time Frame: Week 2 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 39 | 37 | 39 | 38 | 153
units on a scale | -15.9 (15.74) | -17.4 (13.45) | -17.5 (14.61) | -18.2 (14.96) | -17.3 (14.60)

124. Secondary Outcome: Change From Baseline in CDAI at Week 4
Description: CDAI is a composite index for assessing disease activity based on the summation of the counts of TJC28 and SJC28, patient global assessment of disease activity measured on a VAS from 0 to 10 cm, and physician global assessment of disease activity measured on a VAS from 0 to 10 cm. The total CDAI score ranges from 0 to 78 with higher scores indicating higher disease activity. For analysis purposes, all baseline values are defined as the last measurement on or before the first dose of study drug in Study M12-963.
Time Frame: Week 4 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 39 | 157
units on a scale | -20.3 (14.27) | -24.6 (15.61) | -22.1 (13.95) | -24.3 (14.03) | -22.7 (14.43)

125. Secondary Outcome: Change From Baseline in CDAI at Week 6
Description: as for outcome 124
Time Frame: Week 6 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 39 | 157
units on a scale | -25.7 (14.64) | -25.6 (14.71) | -25.8 (13.10) | -25.6 (13.83) | -25.7 (13.95)

126. Secondary Outcome: Change From Baseline in CDAI at Week 8
Description: as for outcome 124
Time Frame: Week 8 of Study M12-963
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 39 | 157
units on a scale | -26.7 (13.68) | -27.0 (13.69) | -28.2 (12.66) | -27.4 (13.92) | -27.3 (13.38)

127. Secondary Outcome: Change From Baseline in CDAI at Week 12
Description: as for outcome 124
Time Frame: Week 12 of Study M12-963 (considered Week 0 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 39 | 157
units on a scale | -28.4 (14.33) | -27.2 (16.72) | -29.7 (12.10) | -28.8 (11.88) | -28.5 (13.76)

128. Secondary Outcome: Change From Baseline in CDAI at Week 16
Description: as for outcome 124
Time Frame: Week 16 (Week 4 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 40 | 35 | 36 | 37 | 148
units on a scale | -28.1 (13.07) | -29.9 (16.04) | -28.5 (12.11) | -29.6 (10.03) | -29.0 (12.84)

129. Secondary Outcome: Change From Baseline in CDAI at Week 20
Description: as for outcome 124
Time Frame: Week 20 (Week 8 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 35 | 38 | 38 | 153
units on a scale | -28.1 (13.05) | -31.8 (14.47) | -28.2 (13.93) | -31.1 (11.44) | -29.7 (13.22)

130. Secondary Outcome: Change From Baseline in CDAI at Week 24
Description: as for outcome 124
Time Frame: Week 24 (Week 12 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 39 | 156
units on a scale | -30.7 (13.81) | -30.1 (15.05) | -28.8 (14.09) | -31.0 (13.15) | -30.1 (13.91)

131. Secondary Outcome: Change From Baseline in CDAI at Week 28
Description: as for outcome 124
Time Frame: Week 28 (Week 16 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 39 | 156
units on a scale | -28.1 (13.27) | -31.4 (15.09) | -29.8 (12.77) | -32.7 (12.79) | -30.4 (13.46)

132. Secondary Outcome: Change From Baseline in CDAI at Week 32
Description: as for outcome 124
Time Frame: Week 32 (Week 20 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 39 | 156
units on a scale | -28.5 (15.08) | -32.4 (14.63) | -29.1 (13.40) | -31.6 (15.08) | -30.3 (14.52)

133. Secondary Outcome: Change From Baseline in CDAI at Week 36
Description: as for outcome 124
Time Frame: Week 36 (Week 24 of Study M12-965)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 39 | 156
units on a scale | -27.6 (14.87) | -30.9 (15.22) | -30.0 (12.28) | -30.9 (14.34) | -29.8 (14.15)

134. Secondary Outcome: Low Disease Activity (LDA) or Clinical Remission (CR) Response Rate Per DAS28 (hsCRP) at Week 2
Description: Percentage of participants achieving LDA or CR on the DAS28 (hsCRP). The DAS28 (hsCRP) is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, hsCRP, and general health are included in the DAS28 (hsCRP) score. Scores range from 0 (no disease activity) to 10 (highest degree of disease activity). LDA was defined as a score from 2.6 to < 3.2, and CR was defined as a score < 2.6. Estimates of the 95% confidence interval of the response rates for each treatment group were calculated using the Agrestil-Coull method.
Time Frame: Week 2 of Study M12-963
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 40 | 37 | 39 | 39 | 155
percentage of participants | 12.5 [5.0 to 26.6] | 8.1 [2.1 to 22.0] | 28.2 [16.4 to 43.9] | 25.6 [14.4 to 41.2] | 18.7 [13.3 to 25.6]

135. Secondary Outcome: LDA or CR Response Rate Per DAS28 (hsCRP) at Week 4
Description: as for outcome 134
Time Frame: Week 4 of Study M12-963
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
percentage of participants | 31.0 [19.0 to 46.1] | 32.4 [19.5 to 48.6] | 30.8 [18.5 to 46.5] | 45.0 [30.7 to 60.2] | 34.8 [27.8 to 42.5]

136. Secondary Outcome: LDA or CR Response Rate Per DAS28 (hsCRP) at Week 6
Description: as for outcome 134
Time Frame: Week 6 of Study M12-963
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
percentage of participants | 45.2 [31.2 to 60.1] | 24.3 [13.2 to 40.3] | 43.6 [29.3 to 59.0] | 50.0 [35.2 to 64.8] | 41.1 [33.8 to 48.9]

137. Secondary Outcome: LDA or CR Response Rate Per DAS28 (hsCRP) at Week 8
Description: as for outcome 134
Time Frame: Week 8 of Study M12-963
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
percentage of participants | 45.2 [31.2 to 60.1] | 27.0 [15.2 to 43.1] | 53.8 [38.6 to 68.4] | 55.0 [39.8 to 69.3] | 45.6 [38.0 to 53.3]

138. Secondary Outcome: LDA or CR Response Rate Per DAS28 (hsCRP) at Week 12
Description: as for outcome 134
Time Frame: Week 12 of Study M12-963 (considered Week 0 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
percentage of participants | 50.0 [35.5 to 64.5] | 35.1 [21.8 to 51.3] | 56.4 [41.0 to 70.7] | 52.5 [37.5 to 67.1] | 48.7 [41.1 to 56.5]

139. Secondary Outcome: LDA or CR Response Rate Per DAS28 (hsCRP) at Week 16
Description: as for outcome 134
Time Frame: Week 16 (Week 4 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 41 | 36 | 37 | 39 | 153
percentage of participants | 51.2 [36.5 to 65.7] | 52.8 [37.0 to 68.0] | 62.2 [46.1 to 76.0] | 48.7 [33.9 to 63.8] | 53.6 [45.7 to 61.3]

140. Secondary Outcome: LDA or CR Response Rate Per DAS28 (hsCRP) at Week 20
Description: as for outcome 134
Time Frame: Week 20 (Week 8 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
percentage of participants | 54.8 [39.9 to 68.8] | 55.6 [39.6 to 70.5] | 56.4 [41.0 to 70.7] | 60.0 [44.6 to 73.7] | 56.7 [48.9 to 64.2]

141. Secondary Outcome: LDA or CR Response Rate Per DAS28 (hsCRP) at Week 24
Description: as for outcome 134
Time Frame: Week 24 (Week 12 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
percentage of participants | 61.9 [46.8 to 75.0] | 44.4 [29.5 to 60.4] | 56.4 [41.0 to 70.7] | 60.0 [44.6 to 73.7] | 56.1 [48.2 to 63.6]

142. Secondary Outcome: LDA or CR Response Rate Per DAS28 (hsCRP) at Week 28
Description: as for outcome 134
Time Frame: Week 28 (Week 16 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
percentage of participants | 47.6 [33.4 to 62.3] | 41.7 [27.1 to 57.8] | 56.4 [41.0 to 70.7] | 55.0 [39.8 to 69.3] | 50.3 [42.6 to 58.0]

143. Secondary Outcome: LDA or CR Response Rate Per DAS28 (hsCRP) at Week 32
Description: as for outcome 134
Time Frame: Week 32 (Week 20 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
percentage of participants | 52.4 [37.7 to 66.6] | 52.8 [37.0 to 68.0] | 61.5 [45.9 to 75.1] | 60.0 [44.6 to 73.7] | 56.7 [48.9 to 64.2]

144. Secondary Outcome: LDA or CR Response Rate Per DAS28 (hsCRP) at Week 36
Description: as for outcome 134
Time Frame: Week 36 (Week 24 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
percentage of participants | 54.8 [39.9 to 68.8] | 41.7 [27.1 to 57.8] | 59.0 [43.4 to 72.9] | 47.5 [32.9 to 62.5] | 51.0 [43.2 to 58.7]

145. Secondary Outcome: CR Response Rate Per DAS28 (hsCRP) at Week 2
Description: Percentage of participants achieving CR on the DAS28 (hsCRP). The DAS28 (hsCRP) is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, hsCRP, and general health are included in the DAS28 (hsCRP) score. Scores range from 0 (no disease activity) to 10 (highest degree of disease activity). LDA was defined as a score from 2.6 to < 3.2, and CR was defined as a score < 2.6. Estimates of the 95% confidence interval of the response rates for each treatment group were calculated using the Agrestil-Coull method.
Time Frame: Week 2 of Study M12-963
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 40 | 37 | 39 | 39 | 155
percentage of participants | 5.0 [0.5 to 17.4] | 5.4 [0.6 to 18.6] | 12.8 [5.1 to 27.2] | 10.3 [3.5 to 24.2] | 8.4 [4.9 to 13.9]

146. Secondary Outcome: CR Response Rate Per DAS28 (hsCRP) at Week 4
Description: as for outcome 145
Time Frame: Week 4 of Study M12-963
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
percentage of participants | 14.3 [6.3 to 28.2] | 8.1 [2.1 to 22.0] | 23.1 [12.4 to 38.5] | 25.0 [14.0 to 40.4] | 17.7 [12.5 to 24.5]

147. Secondary Outcome: CR Response Rate Per DAS28 (hsCRP) at Week 6
Description: as for outcome 145
Time Frame: Week 6 of Study M12-963
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
percentage of participants | 31.0 [19.0 to 46.1] | 18.9 [9.2 to 34.5] | 33.3 [20.6 to 49.1] | 27.5 [16.0 to 43.0] | 27.8 [21.4 to 35.3]

148. Secondary Outcome: CR Response Rate Per DAS28 (hsCRP) at Week 8
Description: as for outcome 145
Time Frame: Week 8 of Study M12-963
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
percentage of participants | 28.6 [17.1 to 43.7] | 21.6 [11.1 to 37.4] | 38.5 [24.9 to 54.1] | 37.5 [24.2 to 53.0] | 31.6 [24.9 to 39.3]

149. Secondary Outcome: CR Response Rate Per DAS28 (hsCRP) at Week 12
Description: as for outcome 145
Time Frame: Week 12 of Study M12-963 (considered Week 0 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
percentage of participants | 31.0 [19.0 to 46.1] | 21.6 [11.1 to 37.4] | 38.5 [24.9 to 54.1] | 40.0 [26.3 to 55.4] | 32.9 [26.1 to 40.6]

150. Secondary Outcome: CR Response Rate Per DAS28 (hsCRP) at Week 16
Description: as for outcome 145
Time Frame: Week 16 (Week 4 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 41 | 36 | 37 | 39 | 153
percentage of participants | 39.0 [25.6 to 54.3] | 30.6 [17.9 to 47.0] | 37.8 [24.0 to 53.9] | 30.8 [18.5 to 46.5] | 34.6 [27.6 to 42.5]

151. Secondary Outcome: CR Response Rate Per DAS28 (hsCRP) at Week 20
Description: as for outcome 145
Time Frame: Week 20 (Week 8 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
percentage of participants | 40.5 [27.0 to 55.5] | 36.1 [22.4 to 52.5] | 25.6 [14.4 to 41.2] | 37.5 [24.2 to 53.0] | 35.0 [28.0 to 42.8]

152. Secondary Outcome: CR Response Rate Per DAS28 (hsCRP) at Week 24
Description: as for outcome 145
Time Frame: Week 24 (Week 12 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
percentage of participants | 33.3 [20.9 to 48.5] | 30.6 [17.9 to 47.0] | 38.5 [24.9 to 54.1] | 45.0 [30.7 to 60.2] | 36.9 [29.8 to 44.7]

153. Secondary Outcome: CR Response Rate Per DAS28 (hsCRP) at Week 28
Description: as for outcome 145
Time Frame: Week 28 (Week 16 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
percentage of participants | 33.3 [20.9 to 48.5] | 27.8 [15.7 to 44.1] | 38.5 [24.9 to 54.1] | 42.5 [28.5 to 57.8] | 35.7 [28.6 to 43.4]

154. Secondary Outcome: CR Response Rate Per DAS28 (hsCRP) at Week 32
Description: as for outcome 145
Time Frame: Week 32 (Week 20 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
percentage of participants | 38.1 [25.0 to 53.2] | 38.9 [24.8 to 55.2] | 35.9 [22.7 to 51.6] | 45.0 [30.7 to 60.2] | 39.5 [32.2 to 47.3]

155. Secondary Outcome: CR Response Rate Per DAS28 (hsCRP) at Week 36
Description: as for outcome 145
Time Frame: Week 36 (Week 24 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
percentage of participants | 38.1 [25.0 to 53.2] | 19.4 [9.4 to 35.3] | 43.6 [29.3 to 59.0] | 37.5 [24.2 to 53.0] | 35.0 [28.0 to 42.8]

156. Secondary Outcome: LDA or CR Response Rate Per CDAI at Week 2
Description: Percentage of participants achieving LDA or CR per CDAI criteria. The CDAI is a composite index for assessing disease activity based on the summation of the counts of TJC28 and SJC28, patient global assessment of disease activity measured on a VAS from 0 to 10 cm, and physician global assessment of disease activity measured on a VAS from 0 to 10 cm. The total CDAI score ranges from 0 to 78 with higher scores indicating higher disease activity. LDA was defined as a score from 2.8 to ≤ 10; CR was defined as a score ≤ 2.8. Estimates of the 95% confidence interval of the response rates for each treatment group were calculated using the Agrestil-Coull method.
Time Frame: Week 2 of Study M12-963
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 39 | 37 | 39 | 39 | 154
percentage of participants | 7.7 [1.9 to 21.0] | 5.4 [0.6 to 18.6] | 12.8 [5.1 to 27.2] | 15.4 [6.9 to 30.1] | 10.4 [6.4 to 16.3]

157. Secondary Outcome: LDA or CR Response Rate Per CDAI at Week 4
Description: as for outcome 156
Time Frame: Week 4 of Study M12-963
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
percentage of participants | 23.8 [13.3 to 38.7] | 21.6 [11.1 to 37.4] | 23.1 [12.4 to 38.5] | 35.0 [22.1 to 50.5] | 25.9 [19.7 to 33.3]

158. Secondary Outcome: LDA or CR Response Rate Per CDAI at Week 6
Description: as for outcome 156
Time Frame: Week 6 of Study M12-963
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
percentage of participants | 40.5 [27.0 to 55.5] | 21.6 [11.1 to 37.4] | 43.6 [29.3 to 59.0] | 45.0 [30.7 to 60.2] | 38.0 [30.8 to 45.7]

159. Secondary Outcome: LDA or CR Response Rate Per CDAI at Week 8
Description: as for outcome 156
Time Frame: Week 8 of Study M12-963
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
percentage of participants | 35.7 [22.9 to 50.9] | 27.0 [15.2 to 43.1] | 46.2 [31.6 to 61.4] | 47.5 [32.9 to 62.5] | 39.2 [32.0 to 47.0]

160. Secondary Outcome: LDA or CR Response Rate Per CDAI at Week 12
Description: as for outcome 156
Time Frame: Week 12 of Study M12-963 (considered Week 0 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
percentage of participants | 40.5 [27.0 to 55.5] | 37.8 [24.0 to 53.9] | 46.2 [31.6 to 61.4] | 50.0 [35.2 to 64.8] | 43.7 [36.2 to 51.5]

161. Secondary Outcome: LDA or CR Response Rate Per CDAI at Week 16
Description: as for outcome 156
Time Frame: Week 16 (Week 4 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 40 | 35 | 36 | 38 | 149
percentage of participants | 47.5 [32.9 to 62.5] | 45.7 [30.5 to 61.8] | 55.6 [39.6 to 70.5] | 50.0 [34.8 to 65.2] | 49.7 [41.7 to 57.6]

162. Secondary Outcome: LDA or CR Response Rate Per CDAI at Week 20
Description: as for outcome 156
Time Frame: Week 20 (Week 8 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 35 | 38 | 39 | 154
percentage of participants | 47.6 [33.4 to 62.3] | 45.7 [30.5 to 61.8] | 36.8 [23.3 to 52.8] | 56.4 [41.0 to 70.7] | 46.8 [39.0 to 54.6]

163. Secondary Outcome: LDA or CR Response Rate Per CDAI at Week 24
Description: as for outcome 156
Time Frame: Week 24 (Week 12 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
percentage of participants | 54.8 [39.9 to 68.8] | 44.4 [29.5 to 60.4] | 43.6 [29.3 to 59.0] | 60.0 [44.6 to 73.7] | 51.0 [43.2 to 58.7]

164. Secondary Outcome: LDA or CR Response Rate Per CDAI at Week 28
Description: as for outcome 156
Time Frame: Week 28 (Week 16 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
percentage of participants | 47.6 [33.4 to 62.3] | 44.4 [29.5 to 60.4] | 48.7 [33.9 to 63.8] | 60.0 [44.6 to 73.7] | 50.3 [42.6 to 58.0]

165. Secondary Outcome: LDA or CR Response Rate Per CDAI at Week 32
Description: as for outcome 156
Time Frame: Week 32 (Week 20 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
percentage of participants | 42.9 [29.1 to 57.8] | 55.6 [39.6 to 70.5] | 51.3 [36.2 to 66.1] | 60.0 [44.6 to 73.7] | 52.2 [44.5 to 59.9]

166. Secondary Outcome: LDA or CR Response Rate Per CDAI at Week 36
Description: as for outcome 156
Time Frame: Week 36 (Week 24 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
percentage of participants | 52.4 [37.7 to 66.6] | 44.4 [29.5 to 60.4] | 59.0 [43.4 to 72.9] | 60.0 [44.6 to 73.7] | 54.1 [46.3 to 61.7]

167. Secondary Outcome: CR Response Rate Per CDAI Criteria at Week 2
Description: Percentage of participants achieving CR per CDAI criteria. The CDAI is a composite index for assessing disease activity based on the summation of the counts of TJC28 and SJC28, patient global assessment of disease activity measured on a VAS from 0 to 10 cm, and physician global assessment of disease activity measured on a VAS from 0 to 10 cm. The total CDAI score ranges from 0 to 78 with higher scores indicating higher disease activity. LDA was defined as a score from 2.8 to ≤ 10; CR was defined as a score ≤ 2.8. Estimates of the 95% confidence interval of the response rates for each treatment group were calculated using the Agrestil-Coull method.
Time Frame: Week 2 of Study M12-963
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 39 | 37 | 39 | 39 | 154
percentage of participants | 0.0 [0.0 to 10.7] | 0.0 [0.0 to 11.2] | 2.6 [0.0 to 14.4] | 0.0 [0.0 to 10.7] | 0.6 [0.0 to 4.0]

168. Secondary Outcome: CR Response Rate Per CDAI Criteria at Week 4
Description: as for outcome 167
Time Frame: Week 4 of Study M12-963
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
percentage of participants | 0.0 [0.0 to 10.0] | 2.7 [0.0 to 15.1] | 5.1 [0.5 to 17.8] | 5.0 [0.5 to 17.4] | 3.2 [1.2 to 7.4]

169. Secondary Outcome: CR Response Rate Per CDAI Criteria at Week 6
Description: as for outcome 167
Time Frame: Week 6 of Study M12-963
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
percentage of participants | 2.4 [0.0 to 13.4] | 0.0 [0.0 to 11.2] | 10.3 [3.5 to 24.2] | 5.0 [0.5 to 17.4] | 4.4 [2.0 to 9.0]

170. Secondary Outcome: CR Response Rate Per CDAI Criteria at Week 8
Description: as for outcome 167
Time Frame: Week 8 of Study M12-963
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
percentage of participants | 4.8 [0.5 to 16.6] | 0.0 [0.0 to 11.2] | 17.9 [8.7 to 33.0] | 17.5 [8.4 to 32.3] | 10.1 [6.2 to 15.9]

171. Secondary Outcome: CR Response Rate Per CDAI Criteria at Week 12
Description: as for outcome 167
Time Frame: Week 12 of Study M12-963 (considered Week 0 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 37 | 39 | 40 | 158
percentage of participants | 7.1 [1.8 to 19.7] | 8.1 [2.1 to 22.0] | 12.8 [5.1 to 27.2] | 12.5 [5.0 to 26.6] | 10.1 [6.2 to 15.9]

172. Secondary Outcome: CR Response Rate Per CDAI Criteria at Week 16
Description: as for outcome 167
Time Frame: Week 16 (Week 4 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 40 | 35 | 36 | 38 | 149
percentage of participants | 7.5 [1.9 to 20.6] | 5.7 [0.6 to 19.6] | 11.1 [3.8 to 25.9] | 15.8 [7.1 to 30.8] | 10.1 [6.1 to 16.0]

173. Secondary Outcome: CR Response Rate Per CDAI Criteria at Week 20
Description: as for outcome 167
Time Frame: Week 20 (Week 8 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 35 | 38 | 39 | 154
percentage of participants | 9.5 [3.2 to 22.6] | 11.4 [3.9 to 26.5] | 15.8 [7.1 to 30.8] | 17.9 [8.7 to 33.0] | 13.6 [9.0 to 20.0]

174. Secondary Outcome: CR Response Rate Per CDAI Criteria at Week 24
Description: Percentage of participants achieving CDAI criteria. The CDAI is a composite index for assessing disease activity based on the summation of the counts of TJC28 and SJC28, patient global assessment of disease activity measured on a VAS from 0 to 10 cm, and physician global assessment of disease activity measured on a VAS from 0 to 10 cm. The total CDAI score ranges from 0 to 78 with higher scores indicating higher disease activity. LDA was defined as a score from 2.8 to ≤ 10; CR was defined as a score ≤ 2.8. Estimates of the 95% confidence interval of the response rates for each treatment group were calculated using the Agrestil-Coull method.
Time Frame: Week 24 (Week 12 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
percentage of participants | 7.1 [1.8 to 19.7] | 5.6 [0.6 to 19.1] | 23.1 [12.4 to 38.5] | 20.0 [10.2 to 35.0] | 14.0 [9.4 to 20.4]

175. Secondary Outcome: CR Response Rate Per CDAI Criteria at Week 28
Description: as for outcome 167
Time Frame: Week 28 (Week 16 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
percentage of participants | 9.5 [3.2 to 22.6] | 5.6 [0.6 to 19.1] | 20.5 [10.5 to 35.8] | 20.0 [10.2 to 35.0] | 14.0 [9.4 to 20.4]

176. Secondary Outcome: CR Response Rate Per CDAI Criteria at Week 32
Description: as for outcome 167
Time Frame: Week 32 (Week 20 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
percentage of participants | 7.1 [1.8 to 19.7] | 5.6 [0.6 to 19.1] | 12.8 [5.1 to 27.2] | 15.0 [6.7 to 29.5] | 10.2 [6.3 to 16.0]

177. Secondary Outcome: CR Response Rate Per CDAI Criteria at Week 36
Description: as for outcome 167
Time Frame: Week 36 (Week 24 of Study M12-965)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Number analyzed (Participants) | 42 | 36 | 39 | 40 | 157
percentage of participants | 9.5 [3.2 to 22.6] | 11.1 [3.8 to 25.9] | 17.9 [8.7 to 33.0] | 15.0 [6.7 to 29.5] | 13.4 [8.8 to 19.7]

ADVERSE EVENTS:
Time Frame: Protocol-related treatment-emergent AEs (TEAEs) and treatment-emergent serious adverse events (TESAEs) were collected from the first dose of study drug in study M12-965 until 70 days after the last dose of study drug (up to 32 weeks).
Description: A protocol-related TEAE or TESAE is defined as any AE with onset or worsening reported by a participant from the first dose of study drug in study M12-965 until 70 days have elapsed following discontinuation of ABT-122 administration. Events were collected whether elicited or spontaneously reported by the participant.
Arm/Group | ADA 40 mg EOW / ABT-122 120 mg EOW | ABT-122 60 mg EOW / 120 mg EOW | ABT-122 120 mg EOW / 120 mg EOW | ABT-122 120 mg EW / 120 mg EOW | All ABT-122 120 mg EOW
Serious Adverse Events (participants affected / at risk) | 0/42 | 1/37 | 5/39 | 0/40 | 6/158
Other Adverse Events (participants affected / at risk) | 17/42 | 14/37 | 16/39 | 14/40 | 61/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ADA 40 mg EOW / ABT-122 120 mg EOW (N=42) | ABT-122 60 mg EOW / 120 mg EOW (N=37) | ABT-122 120 mg EOW / 120 mg EOW (N=39) | ABT-122 120 mg EW / 120 mg EOW (N=40) | All ABT-122 120 mg EOW (N=158)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
ENTEROCOLITIS (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
INFLAMMATION OF WOUND (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
MENORRHAGIA (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ADA 40 mg EOW / ABT-122 120 mg EOW (N=42) | ABT-122 60 mg EOW / 120 mg EOW (N=37) | ABT-122 120 mg EOW / 120 mg EOW (N=39) | ABT-122 120 mg EW / 120 mg EOW (N=40) | All ABT-122 120 mg EOW (N=158)
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
DENTAL CARIES (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
GASTRITIS (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2
NODULE (General disorders) | 0 | 1 | 0 | 0 | 1
HEPATIC STEATOSIS (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
HEPATOBILIARY DISEASE (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
LIVER DISORDER (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1
FOOD ALLERGY (Immune system disorders) | 0 | 0 | 0 | 1 | 1
HYPERSENSITIVITY (Immune system disorders) | 0 | 1 | 0 | 1 | 2
ATYPICAL PNEUMONIA (Infections and infestations) | 1 | 0 | 0 | 0 | 1
BRONCHITIS (Infections and infestations) | 0 | 3 | 0 | 0 | 3
CYSTITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 1
HERPES VIRUS INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 4 | 0 | 0 | 0 | 4
ORAL HERPES (Infections and infestations) | 0 | 0 | 1 | 0 | 1
PARAMETRITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 1
PARONYCHIA (Infections and infestations) | 0 | 0 | 0 | 1 | 1
PHARYNGITIS (Infections and infestations) | 1 | 0 | 0 | 1 | 2
PNEUMONIA (Infections and infestations) | 0 | 0 | 1 | 0 | 1
PULPITIS DENTAL (Infections and infestations) | 1 | 0 | 0 | 0 | 1
RASH PUSTULAR (Infections and infestations) | 1 | 0 | 0 | 0 | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 1
SINUSITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 1
TONSILLITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 3 | 6 | 5 | 15
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1 | 1 | 2
VARICELLA (Infections and infestations) | 0 | 1 | 0 | 0 | 1
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 1
CHEST INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
CONTUSION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
LIMB INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
SKIN ABRASION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
SUBCUTANEOUS HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
THERMAL BURN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
ALANINE AMINOTRANSFERASE ABNORMAL (Investigations) | 1 | 0 | 0 | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 1 | 0 | 2
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 1 | 0 | 2
BLOOD CHOLESTEROL INCREASED (Investigations) | 1 | 0 | 0 | 1 | 2
BLOOD SODIUM DECREASED (Investigations) | 0 | 0 | 1 | 0 | 1
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 1 | 0 | 0 | 1 | 2
EOSINOPHIL COUNT INCREASED (Investigations) | 0 | 0 | 0 | 1 | 1
HAEMOGLOBIN DECREASED (Investigations) | 0 | 0 | 1 | 0 | 1
HEPATIC ENZYME INCREASED (Investigations) | 1 | 0 | 0 | 0 | 1
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 | 1 | 0 | 0 | 1
TRANSAMINASES INCREASED (Investigations) | 0 | 1 | 0 | 0 | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4 | 2 | 9
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 2
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 2
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 3
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 2
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 0 | 4
TENDON DISORDER (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
DIZZINESS (Nervous system disorders) | 0 | 1 | 1 | 0 | 2
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
ADNEXA UTERI CYST (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 1
OVARIAN CYST (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
NAIL DISCOLOURATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
RASH VESICULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
HAEMATOMA (Vascular disorders) | 0 | 0 | 1 | 0 | 1
HYPERTENSION (Vascular disorders) | 0 | 0 | 1 | 1 | 2
VARICOSE VEIN (Vascular disorders) | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.